CLINICAL TRIAL: NCT01507935
Title: Randomised, Controlled, Double-blind Exploratory Study to Investigate the Effect of Specific Prebiotic Oligosaccharides on Gut Microbiota Composition in Healthy Infants
Brief Title: Colonisation Resistance Study
Acronym: ColoR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn due to change of the study product formulation.
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: COL.1.C/A
Record Dates: First submitted 2012-01-05; First posted 2012-01-11 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Healthy Infants
Keywords: Healthy infants; Infant formula; Prebiotics oligosaccharides; Colonisation Resistance; Gut Microbiota

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention Group I (Active Comparator): Healthy infants receiving regular non-hydrolysed cow's milk based infant formula with added prebiotic oligosaccharides mixture I
  Interventions: Other: Regular non-hydrolysed cow's milk
- Intervention Group II (Active Comparator): Healthy infants receiving regular non-hydrolysed cow's milk based infant formula with added prebiotic oligosaccharides mixture II
  Interventions: Other: Regular non-hydrolysed cow's milk
- Control Group (Placebo Comparator): Healthy infants receiving regular non-hydrolysed cow's milk based infant formula with the same composition as the Investigational Formulas but without supplementation of prebiotic oligosaccharides
  Interventions: Other: Regular non-hydrolysed cow's milk
- Reference group (No Intervention): Exclusively breast-fed infants

INTERVENTIONS:
Other: Regular non-hydrolysed cow's milk — Regular non-hydrolysed cow's milk with added prebiotic oligosaccharides mixture I
  Arms: Intervention Group I
Other: Regular non-hydrolysed cow's milk — Regular non-hydrolysed cow's milk with added prebiotic oligosaccharides mixture II
  Arms: Intervention Group II
Other: Regular non-hydrolysed cow's milk — Regular non-hydrolysed cow's milk with the same composition as the Investigational Formulas but without supplementation of prebiotic oligosaccharides
  Arms: Control Group

SUMMARY:
This study is initiated to investigate the effect of infant formulas with added specific prebiotic oligosaccharides on the reduction of specific potential pathogens and/or toxins.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants (gestational age 37 to 42 weeks) aged 2-2.5 months at inclusion
* Fully formula fed for at least one week (not applicable for the breastfeeding reference group since these infants must be exclusively breastfed before and throughout the study)
* Parents' or guardian's written informed consent

Exclusion Criteria:

* Being weaned before inclusion (introduction of any other foods other than formula or breast milk.)
* Moderate or severe acute malnutrition, defined as weight-for-age and sex below -2 z-scores of the median WHO growth standards
* Disorders requiring a special diet (such as food intolerance or food allergy or complaints such as reflux, constipation and cramps)
* Significant congenital abnormality that could affect the study results
* Use of systemic antibiotics or anti-mycotic drugs in the 4 weeks preceding the study
* Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study
* Gastroenteritis in the last two weeks before inclusion

Ages: 8 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition and its metabolic activity | Week 6
  * Gut microbiota composition: count and/or proportion and/or prevalence of group/genus/species of bacteria in the gut
  * Metabolic activity of the gut microbiota: pH, SCFA, lactate

SECONDARY OUTCOMES:
Gastrointestinal symptoms (incidence and severity) | Week 1, Week 3, Week 6, Week 8
Anthropometry | Week 1, Week 3, Week 6, Week 8
Number, type and severity of (serious) adverse events | Week 1, Week 3, Week 6, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Sungkom Jongpiputvanich, A/Prof., MD., Principal Investigator — Chulalongkorn University
Locations (2):
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok